CLINICAL TRIAL: NCT04108221
Title: Randomised Study of Noninferiority Comparing a TransversusAbdominis Plane Block Surgical (c-TAP Block) to the Ultrasound-guided Abdominis Plane Block Transversus (Us-TAP Block) in Postoperative Analgesia After Laparoscopy or Laparotomy
Brief Title: Study Comparing Two Methods of TransversusAbdominis Plane
Acronym: CHIRTAP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator condition
Sponsor: Institut Jean-Godinot (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-A01444-53
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: two arms : arm A : c-TAP Block performed by surgeon arm B : us-TAP Block performed by anesthetist
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : c-TAP Block performed by surgeon (Experimental): c-TAP Block Block performed by surgeon
  Interventions: Procedure: laparoscopy or laparotomy withTransversusAbdominis Plane Block
- Arm B : us-TAP Block performed by anesthetist (Active Comparator): us-TAP Block by anesthetist
  Interventions: Procedure: laparoscopy or laparotomy withTransversusAbdominis Plane Block

INTERVENTIONS:
Procedure: laparoscopy or laparotomy withTransversusAbdominis Plane Block — The US-TAP is performed by the anesthetist under ultrasound control after the end of the procedure of laparoscopy or laparotomy. Under sterile conditions, the anesthetist identifies the oblique abdominal muscles externally, obliquely internally and transversely by ultrasound. A 20 ml needle of 0.5% ropivacaine is injected.
  The surgical TAP (c-TAP) block is performed by the surgeon at the end of the procedure of laparoscopy or laparotomy.The needle and the product used are identical to those of the us-TAP block. The positioning of the needle is in the plane of the fascia between the internal oblique muscle and the transverse muscle, identified by a significant loss of resistance.

SUMMARY:
Interventional, randomised, prospective, multicentric study

DETAILED DESCRIPTION:
Interventional, randomised, prospective, multicentric and single blind study

Primary objective :

demonstrate the equivalence of c-TAP Block to us-TAP Block in postoperative analgesia

Secondary objective :

* Assess the effectiveness of c-TAP block on us-TAP Block in the obese and/or malnourished patient subgroup
* Compare the running time of the c-TAP Block to the us-TAP Block
* Assess the safety of the c-TAP Block gesture in terms of trauma to the intraperitoneal organs by the injection needle two groups:
* Arm A : c-TAP Block performed by the surgeon
* Arm B : us-TAP Block performed by the anesthesist under ultrasound control

Schedule :

* Inclusions start at: 16/09/2019
* End date of inclusions: 31/03/2022
* End date of follow-up: 01/04/2022
* Study report: 30/09/2022

ELIGIBILITY:
Inclusion Criteria:

Patient over 18 years old

* Patient undergoing laparoscopic or laparotomic abdominal surgery at the investigator hospital.
* Patient mastering the French language
* Patient who received informed information about the study and signed a consent
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patients with chronic pain
* Patients with opioid dependence
* Patients allergic to local anesthetic
* Patient who has not signed the consent of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Evolution pain intensity scores, assessed by the numerical pain scale (EN), postoperative and need for systemic analgesics (intravenously or by mouth) during the 24 hours following the end of the procedure | 24 hours
  Evolution pain intensity scores, assessed by the numerical pain scale (EN 1 up to 10)

SECONDARY OUTCOMES:
Failure rate in the obese and / or malnourished patient subgroup | 24 hours
  The failure will be defined as follows: a pain evaluated at> 4/10 on EN that requires intravenous or systemic analgesia
Time in minutes of each of the TAP Block techniques | 24 hours
  The time will be quantified with a stopwatch. For the c-TAP, the stopwatch will be started as soon as the injection equipment of the locoregional anesthesia is received. For the us-TAP block, the stopwatch will be started after the end of the surgical procedure and as soon as the anesthetist starts to wash his hands to proceed with the injection
Occurrence of trauma to the intra-abdominal organs caused by the injection needle | 24 hours
  number of traumas that have occurred

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe EYMARD, PI, Principal Investigator — Institut GODINOT
Locations (1):
- Institut Godinot, Reims, France